CLINICAL TRIAL: NCT00995826
Title: CS-8958 - A Phase I, Double-blind, Placebo-controlled, Ascending, Multiple Dose, Safety, Tolerability and Pharmacokinetic Study in Healthy Subjects.
Brief Title: Safety, Tolerability and Pharmacokinetic Study of Multiple Doses of CS-8958
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biota Scientific Management Pty Ltd (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: Vaxart (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0002; 1UC1AI062373-01 (NIH); 08-0002 (Other Grant/Funding Number: NIAID DMID); 2008-000911-14 (EudraCT Number)
Record Dates: First submitted 2009-10-11; First posted 2009-10-15 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — CS 8958; laninamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Other: Placebo
- CS-8958 DPI (Experimental)
  Interventions: Drug: CS-8958

INTERVENTIONS:
Drug: CS-8958 — Inhaled CS-8958
  Other Names: Laninamivir
  Arms: CS-8958 DPI
Other: Placebo — Inhaled placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to test the safety and tolerability of an investigational multi-dose inhaled flu medication, CS-8958. Study participants will include 16 males and females, aged 18-55 years of age, inclusive. Participants will be divided into two treatment groups (Groups A and B) with each group consisting of 8 subjects. Participants will be involved in study related procedures for a maximum of 14 weeks from initial screen to the follow up visit. 6 subjects in Group A will be administered 40 mg of CS-8958 drug and two subjects will receive placebo (substance containing no medication), once a week for six weeks. In Group B six subjects will be administered 40 mg of CS-8958 drug and two subjects will receive placebo, twice a week for six weeks. Study procedures will include blood and urine samples, ECGs (measure of heart activity), blood pressure, pulse rate and functional oxygen saturation of arterial hemoglobin. Also continuous cardiac telemetry will be performed as well as physical examinations and spirometry assessments.

DETAILED DESCRIPTION:
Influenza is an acute febrile illness caused by influenza A and B virus affecting all age groups.Influenza occurs annually and each year it is estimated that influenza epidemics cause 36,000 deaths and 114,000 hospitalizations in the US alone. Control of human influenza virus infections continues to be a major public health goal.Influenza infects the respiratory tract with a rapid onset of symptoms typically characterized by fever, chills, myalgia, headache, malaise, sore throat and cough. Influenza infections are generally self-limiting; however significant morbidity and mortality can occur, predominantly in high risk groups such as the elderly and those suffering from chronic conditions. It is the objective of this clinical trial to investigate safety and tolerability of multiple doses of CS-8958 administered via inhalation in healthy adult subjects. The pharmacokinetics required for this dosing regimen is only achievable by inhalation delivery. Study participants will include 16 males and females, aged 18-55 years of age, inclusive. The primary objective is to evaluate the safety and tolerability of 40mg CS-8958 once or twice a week (on consecutive days) for 6 weeks in healthy adult subjects after multiple doses administered via inhalation. The secondary objective is to assess the systemic exposure of CS-8958 and its active metabolite R-125489 after single and multiple doses of CS-8958 in healthy adult subjects.

Participants will be divided into two treatment groups (Groups A and B) with each group consisting of 8 subjects. Participants will be involved in study related procedures for a maximum of 14 weeks from initial screen to the follow up visit. 6 subjects in Group A will be administered 40 mg of CS-8958 drug and two subjects will receive placebo (substance containing no medication, once a week for six weeks. In Group B six subjects will be administered 40 mg of CS-8958 drug and two subjects will receive placebo, twice a week for six weeks.

Adverse events will be recorded at every visit. Vital signs including blood pressure, pulse rate and functional oxygen saturation of arterial hemoglobin will be measured on admission, pre-dose and at multiple time points post each dose. ECGs will be performed on admission, pre-dose and at multiple time points post each dose.Continuous cardiac telemetry will be performed for 24 hours post first dose each week for cohort A and 60 hours post first dose each week for cohort B. Spirometry assessments including forced vital capacity, forced expiratory volume in 1 second, forced expiratory volume percentage in 1 second, forced expiratory flow rate, and peak expiratory flow rate will be performed on admission, pre-dose and at multiple time points post dose. Physical examinations will be performed on Day -1 and at the final visit (and as needed if subject develops symptomatology). Blood samples for hematology and biochemistry assessments will be taken on admission, and 24 hours post dose each week. Urine samples for urinalysis tests will be collected on admission, and 24 hours post dose each week. Blood samples for pharmacokinetic testing will be taken pre-dose and at multiple time points post each dose.

The Safety Monitoring Committee (SMC) will review the safety, tolerability and pharmacokinetic data from Cohort A prior to beginning Cohort B.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects aged 18 to 55 years, inclusive

Exclusion Criteria:

* Pregnant or lactating female subjects.
* Out of range findings in vital signs, physical examination, or lab tests.
* Intake of any investigational drug within the 4 months prior to Day 0.
* Positive urine drug screen or alcohol breath test.
* Significant disease, event, or condition which may impact on subject safety or study compliance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be assessed via occurrences of treatment-emergent adverse events, changes in vital signs including BP, PR, SpO2, temperature, ECG, spirometry, physical examinations, and laboratory parameters | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Jane Ryan, PhD, Principal Investigator — Biota Scientific Management Pty Ltd
Locations (1):
- Covance Clinical Research Unit Limited, Leeds, United Kingdom